CLINICAL TRIAL: NCT01558310
Title: A Double - Blind, Placebo Controlled Crossover Study to Evaluate The Efficacy and Tolerability of Stelara ™ (Ustekinumab) in The Treatment of Scalp Psoriasis
Brief Title: A Study to Evaluate the Effectiveness of STELARA ™ (USTEKINUMAB) in the Treatment of Scalp Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Paul Steven Yamauchi, MD, PhD (Individual)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Sponsor-Investigator, Paul Steven Yamauchi, MD, PhD, Medical Director, Clinical Science Institute, Yamauchi, Paul Steven, M.D., Ph.D.
Organization: Yamauchi, Paul Steven, M.D., Ph.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CSI ScalpPsor 012011
Record Dates: First submitted 2012-03-13; First posted 2012-03-20 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Scalp Psoriasis; Plaque Psoriasis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Subjects will be randomized into one of two groups. Group A will receive ustekinumab at week 0, 4, 16, 28, and week 40 and placebo at week 12 and 52.The subjects when assigned to ustekinumab, depending on body weight, will receive either 45mg or 90mg ustekinumab doses
  Interventions: Drug: Ustekinumab; Drug: Placebo
- Group B (Placebo Comparator): Group B will receive placebo at Week 0 and 4, and ustekinumab at weeks 12, 16, 28, 40 and 52. The subjects when assigned to ustekinumab, depending on body weight, will receive either 45mg or 90mg ustekinumab doses
  Interventions: Drug: Ustekinumab; Drug: Placebo

INTERVENTIONS:
Drug: Ustekinumab — Subjects will be randomized into one of two groups. Group A will receive ustekinumab at week 0, 4, 16, 28, and week 40 and placebo at week 12 and 52. Group B will receive placebo at Week 0 and 4, and ustekinumab at weeks 12, 16, 28, 40 and 52. The subjects when assigned to ustekinumab, depending on body weight, will receive either 45mg or 90mg ustekinumab doses
Drug: Placebo — Subjects will be randomized into one of two groups. Group A will receive ustekinumab at week 0, 4, 16, 28, and week 40 and placebo at week 12 and 52. The subjects when assigned to ustekinumab, depending on body weight, will receive either 45mg or 90mg ustekinumab doses

SUMMARY:
This is a single site, randomized, placebo-controlled, cross-over trial of sub-cutaneous injections of placebo and Stelara™ (ustekinumab) in subjects with scalp psoriasis.The purpose of the study is to assess the effectiveness of Stelara™ (ustekinumab)in the treatment of scalp psoriasis by determining the proportion of subjects who clear or almost clear in scalp specific physician assessments. The study will include approximately 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent and the consent must be obtained prior to any study related procedures.
* Be 18 years of age or older at the time of consent; may be male or female.
* Have had a diagnosis of plaque psoriasis at least 6 months prior to administration of study agent.
* Presence of moderate or severe psoriasis on the body other than the scalp.
* At least 30% of scalp affected with erythema, induration and desquamation and s-PGA score greater than or equal to 4.
* Be candidates for phototherapy or systemic treatment of psoriasis.
* Women of childbearing potential and all men must be using adequate birth control measures (eg abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) and must agree to continue use of such measures and not become pregnant or plan a pregnancy until 12 months after receiving the last injection of study agent.
* Be able to adhere to protocol requirements and study visit schedule.
* Must agree not to receive a live virus or live bacterial vaccination during the trial and 12 months after last study injection.
* Must agree not to receive a BCG vaccination during the trial and up to 12 months after the last injection.
* Must avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during the study.
* Are considered eligible according to the following tuberculosis (TB) screening criteria:

  * Have no history of latent or active TB prior to screening. An exception is made for subjects currently receiving treatment for latent TB with no evidence of active TB, or who have a history of latent TB and documentation of having completed appropriate treatment for latent TB within 3 years prior to the first administration of study agent. It is the responsibility of the investigator to verify the adequacy of previous antituberculous treatment and provide appropriate documentation.
  * Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
  * Within 6 weeks prior to the first administration of study agent, have a negative QuantiFERON-TB Gold test result (see Attachment #).Indeterminate results should be handled as outlined in Section #, Exclusion Criteria.
  * Have a chest radiograph (both posterior-anterior and lateral views), taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current, active TB or old, inactive TB.
* Have screening laboratory test results within the following parameters:

  * Hemoglobin > 10g/dL
  * White Blood Cells > 3.5 x 109 /L
  * Neutrophils > 1.5 x 109 /L
  * Platelets > 100 X109 /L
  * Serum Creatinine < 1.5 mg/dL ( or 133 micromol/L )
  * AST,ALT, and alkaline phosphatase levels must be within 1.5 times the upper limit of normal range for the laboratory conducting the test

Exclusion Criteria:

Subjects meeting any of the following criteria may not be enrolled in the study:

* Currently have non-plaque forms of psoriasis (erythrodermic, guttate, or pustular).
* Have current drug-induced psoriasis.
* Presence of any skin conditions ( including scalp) other than psoriasis that would interfere with evaluations of the effect of study agents.
* Are pregnant, nursing, or planning pregnancy (both men and women) while enrolled in the study.
* Have used any therapeutic agent targeted at reducing IL-12 and/or IL-23, including but not limited to ustekinumab and ABT -874.
* Have used any investigational drug within the previous 4 weeks or 5 times the half-life of the investigational agent, whatever is longer.
* Have used any investigational drug within the previous 3 months or 5 times the half-life of the biological, whichever is longer.
* Have ever received natalizumab or other agents that target alpha-4-integrin.
* Have received phototherapy or any any systemic medications/treatments that could affect psoriasis or s-PGA/PASI evaluations ( including but not limited to, oral or injectable corticosteroids, retinoids,1,25 dihydroxy vitamin D3 and analogues, psoralens, sulfasalazine, hydroxyurea, or fumaric acid derivatives) within 4 weeks of administration of study agent.
* Have used topical mediations/treatments that could affect psoriasis or s-PGA/PASI evaluation ( eg corticosteroids , anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen,trimethylpsoralens) within 2 weeks of the first administration of study agent.
* Have used any systemic immunosuppressants ( eg Methotrexate, azathioprine, cyclosporine,6-thioguanine, mercaptopurine, mycophenolate, mofetil, hydroxyurea, and tacrolimus) within 4 weeks of the first administration of study agent.
* Are currently receiving lithium, anti-malarials, or intramuscular gold, or have received lithium, anti-malarials, or intramuscular gold, or have received lithium, anti-malarials, or intramuscular gold within 4 weeks of the first administration of study agent.
* Have received within 3 months prior to the first injection a live virus or bacterial vaccination. Subjects must agree not to receive a live virus or bacterial vaccination during the trial or up to 12 month after the last study agent injection.
* Have had a BCG vaccination within 12 months of screening. Subject must agree not to receive a BCG vaccination during the trial or up to 12 months after the last study agent injection.
* Have a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infections (eg bronchiectasis), recurrent urinary tract infections (recurrent pyelonephritis or chronic non-remitting cystitis), or open, draining, or infected skin wounds or ulcers.
* Have or have had a serious infection (eg sepsis, pneumonia,or pyelonephritis) or have been hospitalized or received IV antibiotics for an infection during the 2 months prior to screening
* Have a history of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, prior to screening.
* Have persistently indeterminate (indeterminate on repeat sampling) QuantiFERON-TB Gold test results
* Have had a Bacille Calmette-Guérin (BCG) vaccination within 12 months of screening.
* Have a chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of a malignancy or current active infection, including TB.
* Have had a non-tuberculous mycobacterial infection or opportunistic infection (eg, cytomegalovirus, pneumocystosis, aspergillosis) within 6 months prior to screening.
* Known to be infected with human immunodeficiency virus, hepatitis B, or hepatitis C.
* Have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease.
* Have a transplanted organ.
* Have a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and /or splenomegaly.
* Have a known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin or cervix that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to the first administration of study agent).
* Have been hospitalized in the past 3 years for asthma, ever required intubation for treatment of asthma, currently require oral corticosteroids for the treatment of asthma, or required more than one short -term (< 2 weeks) course of oral corticosteroids for asthma within the previous year.
* Have undergone allergy immunotherapy previously for prevention of anaphylactic reactions.
* Have shown a previous immediate hypersensitivity response, including anaphylaxis, to an immunoglobulin product (eg plasma derived or recombinant monoclonal antibody).
* Be known to have had a substance abuse (drug or alcohol) problem within the previous 12 months.
* Be participating in another trial using an investigational agent or procedure during participation in the trial.
* Use of tar shampoos within 14 days of first dose of study drug.
* Use of OTC shampoos for scalp psoriasis will not be allowed during study.
* Use of topical corticosteroids or other topical agents for the treatment of psoriasis on the scalp will not be allowed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
s-PGA ( Scalp specific Physician Global Assessment) at Week 12 | Week 12 (8 weeks after the second of two SC doses of ustekinumab)
  s-PGA (Scalp specific Physician Global Assessment) is a 7 point scale ranging from 0 (Clear = No signs of psoriasis ) to 6 (Severe = Very marked plaque elevation, scaling, and/or erythema)

CONTACTS AND LOCATIONS:
Overall Officials: PAUL S YAMAUCHI, MD,PhD, Principal Investigator — Clinical Science Institute
Locations (1):
- Clinical Science Institute, Santa Monica, California, United States